CLINICAL TRIAL: NCT01057082
Title: Dietary Supplements and Aging Muscle: Specific Amino Acids to Combat Sarcopenia
Brief Title: Dietary Supplements and Aging Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Amy Ellis, Registered Dietitian; Graduate Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F100107001; F31AT005384-01 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Aging; Muscle; Dietary Supplement; HMB; Arginine; Glutamine
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Juven (Experimental): Participants in the treatment arm will receive the dietary supplement Juven.
  Interventions: Dietary Supplement: Juven
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Juven

INTERVENTIONS:
Dietary Supplement: Juven — Participants in the treatment arm will be asked to consume 2 packets of Juven drink mix each day for a period of six months.
  Arms: Juven
Dietary Supplement: Juven — Participants in the placebo arm will be asked to consume two packets of an orange-flavored drink mix each day for a period of six months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether older adults (ages 65-89) who consume the dietary supplement Juven (Abbott Laboratories) versus placebo for 6 months will demonstrate increases in fat-free mass, muscle volume,and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 65-89
* Ambulatory

Exclusion Criteria:

* Cognitive impairment
* History of renal or hepatic disease
* History of hypotension
* History of peripheral artery disease
* Uncontrolled hypertension
* Uncontrolled diabetes
* Self-reported claustrophobia
* Current smoker
* Steroid or androgen use with the previous 3 months
* Individuals with pacemakers and defibrillators

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fat-free mass as determined by a four-compartment model of body composition | Baseline, 3-months, 6-months

SECONDARY OUTCOMES:
Appendicular lean mass as determined by dual energy X-ray absorptiometry | Baseline, 3-months, 6-months
Muscle volume as determined by magnetic resonance imaging | Baseline and 6-months
Physical function as determined by questionnaire and a battery of physical performance tests | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Ellis, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ellis AC, Hunter GR, Goss AM, Gower BA. Oral Supplementation with Beta-Hydroxy-Beta-Methylbutyrate, Arginine, and Glutamine Improves Lean Body Mass in Healthy Older Adults. J Diet Suppl. 2019;16(3):281-293. doi: 10.1080/19390211.2018.1454568. Epub 2018 Apr 19. PMID 29672184